CLINICAL TRIAL: NCT01814592
Title: Comparison of Two Bilaminar Techniques for Root Covering of Miller´s Recessions Class I and II: A Blind, Randomized Controlled Clinical Trial
Brief Title: Comparison Between Two Coronally Positioned Flap With Connective Tissue
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Universidad El Bosque, Bogotá (Other)
Responsible Party: Principal Investigator, Sergio Iván Losada Amaya, Professor, DDS, specialist in periodontics and oral medicine, Universidad El Bosque, Bogotá
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PCI-2012-359
Record Dates: First submitted 2013-03-11; First posted 2013-03-20 (Estimated); Last update posted 2013-03-26 (Estimated); Status verified 2013-03

CONDITIONS: Gingival Recession; Periodontal Atrophy
Keywords: coronally positioned flap; connective tissue; gingival margin; gingival recession/ treatment; gingival recession/ surgery; subepithelial connective tissue graft; randomized controlled clinical trial; surgical flaps; Treatment outcome
MeSH Terms: conditions — Gingival Recession; Periodontal Atrophy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- coronally mucosal thickness flap (Experimental): coronally mucosal thickness flap plus connective tissue graft for root coverage (subepithelial connective tissue graft)
  Interventions: Procedure: coronally mucosal thickness flap
- coronally partial thickness flap (Active Comparator): coronally partial thickness flap plus connective tissue for root coverage (subepithelial connective tissue graft)
  Interventions: Procedure: coronally partial thickness flap plus connective tissue

INTERVENTIONS:
Procedure: coronally partial thickness flap plus connective tissue — The design of the flap will be performed according to the technique described by de Sanctis and Zucchelli 2007.
  Other Names: subepithelial connective tissue graft; coronally positioned flap
  Arms: coronally partial thickness flap
Procedure: coronally mucosal thickness flap — The design of the flap will be performed according to the technique described by Greenwell H, Vance G, Munninger B and Johnston H.
  Other Names: superficial-layer split-tihickness flap
  Arms: coronally mucosal thickness flap

SUMMARY:
The aim of this study is to evaluate the effectiveness of total root coverage between two coronally positioned flap technique in Miller recession Class I and II, in patients attending at "Universidad El Bosque" dental school clinics.

DETAILED DESCRIPTION:
This is a blind, randomized controlled clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Class I and II Miller recessions showing a recession depth ≥ 2 mm.
* Recessions isolated and / or maximum continuous two teeth.
* Recessions in incisors, canines and premolars
* Patients 20 to 60 years old.

Exclusion Criteria:

* Systemic compromise, that contraindicates any periodontal surgical procedure.

  * Warfarin medication.
  * Uncontrolled diabetes mellitus with glycosylated hemoglobin ≥ 8
  * Chronic steroid therapy (dose of 7.5 mg/ day for more than 14 days)
  * HIV-AIDS infection with CD4 counts <200.
  * Immunosuppression.
* Recessions molars not be taken into account in the study.
* Patients who have used antibiotics one month prior to the surgical procedure.
* Pregnancy.
* Active smoker.
* Patients with a history of periodontal surgery at the recession area that has taken place in the last three months.
* Severe dental malposition, teeth rotation, versions teeth root coverage that contraindicates surgery.
* Non carious cervical lesions or caries where is not visible the cemento- enamel junction (CEJ).
* Active inflammation that contraindicates surgical procedure of the recession.
* Active Orthodontics

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2013-03; Primary Completion 2014-04 (Estimated); Study Completion 2014-08 (Estimated)

PRIMARY OUTCOMES:
Assess percentage of total root coverage between two subepithelial conective tissue graft technique for covering Class I and II Miller recessions patients attending at dental clinics of "Universidad El Bosque" | one month (plus or minus 2 days), three months (plus or minus 3 days) and six months (plus or minus 5 days)

SECONDARY OUTCOMES:
Assess the proportion of root coverage | one month (plus or minus 2 days), Three months (plus or minus 3 days) and six month (plus or minus 5 days)
Clinical attachment level, width of keratinized tissue and the position of the mucogingival junction following root coverage procedures | one month (plus or minus 2 days), three months (plus or minus 3 days) and six months (plus or minus 5 days)

OTHER OUTCOMES:
Assess the frequency of adverse events | 0 hours (intrasurgical), 1-24 hours (immediate postoperative), 25 hours to 6 days (mediate postoperative) and 7 or more days (late postoperative)

CONTACTS AND LOCATIONS:
Overall Officials: Sergio I Losada Amaya, Professor, Principal Investigator — Universidad El bosque- UNIECLO; Jaime A Marquez Cristo, Professor, Study Chair — Universidad El Bosque- UNIECLO; Miguel F Vargas del Campo, Professor, Study Chair — Universidad El Bosque- UNIECLO; Silie S Arboleda Salaiman, Professor, Study Chair — Universidad El Bosque- UNIECLO; Maria I Pardo Silva, Professor, Study Director — Universidad El Bosque- UNIECLO
Locations (1):
- Universidad El Bosque, Bogotá, D. C., Bogotá, D. C., Colombia